CLINICAL TRIAL: NCT05452616
Title: Same-day Versus Rapid ART Initiation in HIV-positive Individuals Presenting With Symptoms of Tuberculosis: an Open-label Randomized Non-inferiority Trial in Lesotho and Blantyre District, Malawi
Brief Title: Same-day Versus Rapid ART Initiation in HIV-positive Individuals Presenting With Symptoms of Tuberculosis
Acronym: SaDAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); SolidarMed (Other); Kamuzu University of Health Sciences, Malawi (Unknown); Swiss Tropical & Public Health Institute (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AO_2022-00031; am22Labhardt
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: Tuberculosis (TB) infection; Acquired immunodeficiency syndrome; Antiretroviral therapy (ART); Immune reconstitution inflammatory syndrome; People living with HIV (PLHIV); Same-day initiation (SDI) of ART; TB preventive treatment; Sub-Saharan African countries; HIV/TB-coinfection; immune reconstitution inflammatory syndrome (IRIS)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis; Infections; Immune Reconstitution Inflammatory Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, open-label, 1:1 individually randomized, non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "ART first" arm (Active Comparator): ART initiation on the day of enrolment independent of TB investigations
  Interventions: Other: ART first- Therapeutic use trial
- "TB results first" arm (Active Comparator): ART initiation only after active TB has been refuted or confirmed
  Interventions: Other: TB results first- Therapeutic use trial

INTERVENTIONS:
Other: ART first- Therapeutic use trial — ART initiation on the day of enrolment independent of TB investigations in PLHIV with presumptive TB but no signs of CNS disease. The trial uses treatments and drug-doses as per international and national guidelines. All treatment components will be applied at standard dosage and no new substances or alternative indications will be tested.
  Arms: "ART first" arm
Other: TB results first- Therapeutic use trial — Deferral of ART initiation until active TB has been refuted or confirmed. PLHIV presenting with symptoms (cough, fever, night sweat, weight loss) are defined as presumptive TB, and should have microbiological TB investigations. Routine TB investigations in Malawi and Lesotho usually consist of two sputum bottles for analysis using nucleic acid amplification tests (Xpert MTB/RIF (Ultra)).The trial uses treatments and drug-doses as per international and national guidelines. All treatment components will be applied at standard dosage and no new substances or alternative indications will be tested.
  Arms: "TB results first" arm

SUMMARY:
SaDAPT is a pragmatic, randomized, therapeutic-use trial comparing two approaches ("ART first" versus "TB results first") for the timing of ART initiation in PLHIV with presumptive TB, but no signs of central nervous system (CNS) disease, in a routine primary and secondary care setting in southern Africa with regard to HIV viral suppression (VL <400 copies/mL) 26 weeks after enrolment.

DETAILED DESCRIPTION:
In this randomized controlled trial (RCT) two different, guideline-approved algorithms for antiretroviral therapy (ART) initiation in people living with HIV (PLHIV) with presumptive Tuberculosis (TB), but no signs of central nervous system (CNS) disease will be compared. In one arm, same-day initiation (SDI) of ART will be applied ("ART first") for all participants independent of the status or results of initial TB investigations. In the other arm, an approach with deferral of ART initiation until TB is excluded or confirmed and TB treatment initiated will be applied ("TB results first"). The direct comparison of the two approaches in a pragmatic, two-country RCT conducted in a representative high-prevalence setting will provide evidence on the open question of optimal timing of ART initiation in the large subgroup of PLHIV with presumptive TB outside the CNS.

ELIGIBILITY:
Inclusion Criteria:

* 12 years or older
* HIV-positive
* Not taking ART (naïve or reported no ART intake since 90 days or more)
* Presenting with one or more TB symptoms according to W4SS
* Unknown TB status
* Planning to continue care at the study facility for at least 30 weeks
* Willing and able to consent (age 18 years or older) or assent with guardian consent (age 12 to 17 years)

Exclusion Criteria:

* Medical condition requiring admission or referral to a higher level health facility at enrolment
* Symptoms or clinical signs suggestive for diseases of the CNS
* Positive cryptococcal antigen test (CrAg)
* Reporting to be pregnant
* Taking TB treatment, TB preventive therapy (TPT) or treatment against cryptococcal meningitis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
HIV viral suppression <400 copies/mL | 26 (22 - 40) weeks after enrolment
  HIV viral suppression <400 copies/mL (obtained from routine laboratory reports at study facility, from laboratory reports of referral facility in case of transfer out, or from dried blood spot (DBS) sample for participants without documented clinic visit but found during home visit tracing)

SECONDARY OUTCOMES:
Retention in care | 26 (22 - 30) weeks after enrolment
  Retention in care, defined as a documented ART clinic visit between 22 and 30 weeks after enrolment
Engagement in care | 26 (22 - 30) weeks after enrolment
  Engagement in care, defined as reporting regular ART intake, irrespective if a documented visit took place between 22 and 30 weeks after enrolment
Disengagement from care | 26 (22 - 30) weeks after enrolment
  Disengagement from care, defined as non-engaged in care but reached through patient tracing
Lost to follow-up | 26 (22 - 30) weeks after enrolment
  Lost to follow-up, defined as non-retained in care and not reached through tracing
Non-traumatic mortality | during the first 30 weeks after enrolment
  Non-traumatic mortality
Serious adverse events (SAEs) | during the first 30 weeks after enrolment
  SAEs
TB-Immune reconstitution inflammatory syndrome (IRIS) | during the first 30 weeks after enrolment
  TB-Immune reconstitution inflammatory syndrome (IRIS) is defined as Adverse event of special interest (AESIs): AESIs
Incidence of TB disease (microbiologically confirmed and/or clinical diagnosis) | during the first 30 weeks after enrolment
  Incidence of TB disease (microbiologically confirmed and/or clinical diagnosis), defined as any TB diagnosis after enrolment not classified as prevalent TB at enrolment
HIV viral suppression | at 26 (22 - 40) weeks
  HIV viral suppression using different thresholds (<20 copies/mL; <100 copies/mL; <1000 copies/mL)

OTHER OUTCOMES:
Prevalence of active TB diagnosed at enrolment (exploratory endpoint) | up to a maximum of 28 days after enrolment
  Prevalence of active TB, defined as TB diagnosed clinically or microbiologically through the TB investigations at enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, Prof. Dr. DTM&H, MIH, Principal Investigator — Division of Clinical Epidemiology, University Hospital Basel; Rachael Mary Burke, BMBCh, MSc, DTM&H, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- SolidarMed Lesotho, Premium House #224, Kingsway, Maseru West, Maseru, Lesotho
- Kamuzu University of Health Sciences, Helse Nord Tuberculosis Initiative, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
* An anonymized key dataset necessary for reproducing the primary and key secondary endpoints will be made freely available in an appropriate repository, such as zenodo.org, alongside the publication of the study results. Besides removal of variables not required for key analysis, we will remove participant identifier, study site and exact date information. Requests for access to more detailed data may be made to the corresponding author by submitting a proposal, which will be reviewed by the trial consortium.
  * The statistical report for the primary and key secondary endpoints and the code to produce it will be published together with the data set.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: • Within 3 months after publication of primary results
Access Criteria: • Open access

REFERENCES:
- [Derived] Gerber F, Semphere R, Lukau B, Mahlatsi P, Mtenga T, Lee T, Kohler M, Glass TR, Amstutz A, Molatelle M, MacPherson P, Marake NB, Nliwasa M, Ayakaka I, Burke R, Labhardt N. Same-day versus rapid ART initiation in HIV-positive individuals presenting with symptoms of tuberculosis: Protocol for an open-label randomized non-inferiority trial in Lesotho and Malawi. PLoS One. 2024 Feb 8;19(2):e0288944. doi: 10.1371/journal.pone.0288944. eCollection 2024. PMID 38330045

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT05452616/Prot_002.pdf
  • Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT05452616/SAP_004.pdf